CLINICAL TRIAL: NCT03411798
Title: Sequential Application of Yisaipu® and Disease Modifying Anti-Rheumatic Drugs (DMARDs) in Treating Mild-to-Moderate Ankylosing Spondylitis: the Mid-term Follow-up Result
Brief Title: Sequential Application of Yisaipu® and DMARDs in Treating Mild-to-Moderate AS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-201711-K6
Record Dates: First submitted 2017-12-14; First posted 2018-01-26 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-07

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis(AS); TNFi; Yisaipu®; Disease modifying anti-rheumatic drugs (DMARDs)
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Methotrexate; Sulfasalazine; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Yisaipu® was introduced only during the active state and was switched to DMARDs, methotrexate(MTX), sulfasalazine(SSZ) and hydroxychloroquine(HCQ), after disease remission (ESR & CRP reduce to normal and BASDAI<4) maintenance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Yisaipu® was introduced only during the active state and was switched to DMARDs, methotrexate(MTX), sulfasalazine(SSZ) and hydroxychloroquine(HCQ), after disease remission (ESR & CRP reduce to normal and BASDAI<4) maintenance.
  Interventions: Drug: Yisaipu®

INTERVENTIONS:
Drug: Yisaipu® — Yisaipu® was introduced only during the active state and was switched to DMARDs, methotrexate(MTX), sulfasalazine(SSZ) and hydroxychloroquine(HCQ), after disease remission (ESR & CRP reduce to normal and BASDAI<4) maintenance.
  Other Names: methotrexate(MTX); sulfasalazine(SSZ); hydroxychloroquine(HCQ)

SUMMARY:
The drug regimes in treating ankylosing spondylitis(AS) have limitations. The tumor necrosis factor inhibitors(TNFi) was effective but expensive. Disease modifying anti-rheumatic drugs (DMARDs) were cheap but insufficient. This study proposed a sequential usage of TNFi, the Yisaipu®, and DMARDs, and aims to evaluate the mid-term therapeutic effect of this new scheme in treating the mild-to-moderate AS.

ELIGIBILITY:
Inclusion Criteria:

* 1.Clinical diagnosis of Ankylosing Spondylitis(AS) based on modified New York diagnostic criteria for AS (1984) 2.At the mild-to-moderate stage of AS disease 3.At the active phase of AS disease

Exclusion Criteria:

* 1.Active tuberculosis, hepatitis, tumors, infection diseases or combine with other rheumaimmune systemic diseases or osteoarthritis diseases 2.Pregnant or breastfeeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
ASAS 20 | 3 months after
  Improvement of >20% and >1 unit in at least 3 domains on a scale of 10;No worsening of >20% and >1 unit in remaining domain on a scale of 10 compare to the baseline status
ASAS 20 | 6 months after
  Improvement of >20% and >1 unit in at least 3 domains on a scale of 10;No worsening of >20% and >1 unit in remaining domain on a scale of 10 compare to the baseline status
ASAS 20 | 12 months after
  Improvement of >20% and >1 unit in at least 3 domains on a scale of 10;No worsening of >20% and >1 unit in remaining domain on a scale of 10 compare to the baseline status
ASAS 40 | 3 months after
  Improvement of >40% and >2 unit in at least 3 domains on a scale of 10;No worsening at all in remaining domain compare to the baseline status
ASAS 40 | 6 months after
  Improvement of >40% and >2 unit in at least 3 domains on a scale of 10;No worsening at all in remaining domain compare to the baseline status
ASAS 40 | 12 months after
  Improvement of >40% and >2 unit in at least 3 domains on a scale of 10;No worsening at all in remaining domain compare to the baseline status

SECONDARY OUTCOMES:
BASDAI | baseline,3 months after,6 months after,12 months after
  Bath Ankylosing Spondylitis Disease Activity Index
BASFI | baseline,3 months after,6 months after,12 months after
  BASDAI Bath Ankylosing Spondylitis Functional Index
Patient Global Assessment | baseline,3 months after,6 months after,12 months after
  Measuring disease activity by using the visual analogue scales (VAS) on which patients rated the severity of their symptoms from 0 (none) to 10 (most severe) .
CRP | baseline,3 months after,6 months after,12 months after
  acute-phase reactant(C-reactive protein)
ESR | baseline,3 months after,6 months after,12 months after
  acute-phase reactant(Erythrocyte Sedimentation rate )
SQOL-AS | baseline,3 months after,6 months after,12 months after
  SQOL-AS(The Scale of Quality of Life for Ankylosing Spondylitis) questionnaire consists of physiological function, psychological state, social adaptation and self-awareness 4 dimensions. There are 5 to 8 questions in every dimension. The score ranges are 8 to 40 for physiological function, 6 to 30 for psychological state, 5 to 25 for social adaptation and 6 to 30 for self-awareness. The more score that patients got means the better state they were in that dimension, namely, the batter quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided